CLINICAL TRIAL: NCT03106415
Title: Phase I/II Trial of Pembrolizumab in Combination With Binimetinib in Unresectable Locally Advanced or Metastatic Triple Negative Breast Cancer
Brief Title: Pembrolizumab and Binimetinib in Treating Patients With Locally Advanced or Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1632; NCI-2017-00496 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-009051 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-04-03; First posted 2017-04-10 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-10

CONDITIONS: Breast Adenocarcinoma; Metastatic Triple-Negative Breast Carcinoma; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — binimetinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (binimetinib, pembrolizumab) (Experimental): Patients receive binimetinib PO BID on days 1-14 of cycle 1 and on days 1-21 of cycle 2 and subsequent cycles. Beginning cycle 2, patients also receive pembrolizumab IV over 30 minutes on day 1. Cycle 1 equals 14 days. Cycles 2 and beyond repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162; Mektovi
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I/II trial studies the best dose of pembrolizumab and binimetinib and how well it works when given together with pembrolizumab in treating patients with triple negative breast cancer that has spread to other parts of the body (metastatic). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Binimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab and binimetinib may work better in treating patients with triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of binimetinib in combination with pembrolizumab. (Phase I) II. To evaluate the objective response rate (ORR) of binimetinib in combination with pembrolizumab in patients with unresectable locally advanced or metastatic triple negative breast cancer by Response Evaluation Criteria in Solid Tumors (RECIST). (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of binimetinib in combination with pembrolizumab.

II. To evaluate the ORR by immune-related RECIST criteria (irRECIST). III. To evaluate the progression free survival (PFS), duration of response (DoR), and disease control rate (DCR) by RECIST and irRECIST.

IV. To assess overall survival (OS).

CORRELATIVE RESEARCH OBJECTIVES:

I. To assess the correlation between ORR, PFS, or OS and baseline and/or change in tumor infiltrating lymphocytes (TILs).

II. To assess the correlation between ORR, PFS, or OS and baseline and/or change in immune related gene signature and PDJ amplification.

III. To assess the change in immunoregulatory cells (IRC). IV. To assess the change in the cytokine profile. V. To assess the change in circulating tumor cells (CTC).

OUTLINE: This is phase I, dose-escalation study of binimetinib followed by a phase II study.

Patients receive binimetinib orally (PO) twice daily (BID) on days 1-14 of cycle 1 and on days 1-21 of cycle 2 and subsequent cycles. Beginning cycle 2, patients also receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycle 1 equals 14 days. Cycles 2 and beyond repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months until progressive disease, then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of adenocarcinoma of the breast
* Estrogen receptor (ER) and progesterone receptor (PR) negative; defined as ER =< 10% and PR =< 10% staining by immunohistochemistry (IHC)
* HER2 negative in the primary or metastatic tumor tissue defined as:

  * Immunohistochemistry (IHC) grade 0 as defined by no staining observed or membrane staining that is incomplete and is faint/barely perceptible and within =< 10% of the invasive tumor cell; OR
  * IHC 1+ as defined by incomplete membrane staining that is faint/barely perceptible and within > 10% of the invasive tumor cell; OR
  * IHC grade 2+ staining intensity by means of IHC analysis with no gene amplification below; OR
  * No gene amplification on in situ hybridization (ISH) based on:

    * Single-probe average HER2 copy number < 4.0 signals/cell OR
    * Dual-probe HER2/CEP17 ratio < 2.0 with an average HER2 copy number < 4.0 signals/cell
* For phase II part of the trial: =< 3 prior lines of treatment in the metastatic setting for the current breast cancer; however, there is no limit on number of prior line of therapy in phase I part of the trial
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Hemoglobin >= 9.0 g/dL (must be >= 7 days after most recent transfusion) (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 or >= 1.5 x 10^9/L (obtained =< 14 days prior to registration)
* Platelet count >= 100,000/mm^3 or >= 100 x 10^9/L (must be >= 7 days after most recent transfusion) (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Aspartate transaminase (AST) and/or alanine transaminase (ALT) =< 2.5 x ULN or =< 5 x ULN for patients with liver metastases (obtained =< 14 days prior to registration)
* Creatinine =< 1.5 x ULN OR calculated creatinine clearance must be >= 50 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* International normalized ratio (INR) or prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (obtained =< 14 days prior to registration)
* Adequate cardiac function:

  * Left ventricular ejection fraction (LVEF) >= 50% as determined by multigated acquisition (MUGA) scan or echocardiogram (echo)
  * Corrected QT (QTc) interval =< 480 ms
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Able to swallow oral medication
* Both female and male patients of reproductive potential must agree to avoid pregnancy or impregnating a partner (respectively) while receiving drug and for 120 days after last dose of study drug
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide mandatory tissue and blood for correlative research purposes
* RETREATMENT REGISTRATION: Treatment cannot begin prior to registering to the retreatment phase and will ideally begin =< 7 days after registration for the retreatment phase
* RETREATMENT REGISTRATION: Stopped initial treatment with pembrolizumab and binimetinib after attaining an investigator-determined confirmed complete response (CR) according to RECIST 1.1, and:

  * Was treated for at least 24 weeks with pembrolizumab and binimetinib before discontinuing therapy
  * Received at least 2 cycles with pembrolizumab and binimetinib beyond the date when the initial CR was declared OR
  * Had stable disease (SD), partial response (PR), or CR and stopped pembrolizumab and binimetinib treatment after 24 months of study therapy for reasons other than disease progression or intolerability
* RETREATMENT REGISTRATION: ECOG performance status (PS) 0 or 1
* RETREATMENT REGISTRATION: Hemoglobin >= 9.0 g/dL (must be >= 7 days after most recent transfusion) (obtained =< 14 days prior to re-registration)
* RETREATMENT REGISTRATION: Absolute neutrophil count (ANC) >= 1500/mm^3 or >= 1.5 X 10^9/L (obtained =< 14 days prior to re-registration)
* RETREATMENT REGISTRATION: Platelet count >= 100,000/mm^3 or >= 100 X 10^9/L (must be >= 7 days after most recent transfusion) (obtained =< 14 days prior to re-registration)
* RETREATMENT REGISTRATION: Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to re-registration)
* RETREATMENT REGISTRATION: Aspartate transaminase (AST) and alanine transaminase (ALT) =< 2.5 x ULN or =< 5 x ULN for patients with liver metastases (obtained =< 14 days prior to re-registration)
* RETREATMENT REGISTRATION: Creatinine =< 1.5 x ULN OR calculated creatinine clearance must be >= 50 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to re-registration)
* RETREATMENT REGISTRATION: International normalized ratio (INR) or prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (obtained =< 14 days prior to re-registration)
* RETREATMENT REGISTRATION: Females of childbearing potential should have a negative serum or urine pregnancy test =< 72 hours prior to re-registration
* RETREATMENT REGISTRATION: Females or males of childbearing potential must be willing to use adequate methods of contraception or abstain from heterosexual activity for the course of the study through 120 days after last dose of study medication
* RETREATMENT REGISTRATION: Experienced an investigator-determined confirmed radiographic disease progression after stopping their initial treatment with pembrolizumab and binimetinib

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm OR participated in a study of an investigational agent, received study therapy or used an investigational device =< 4 weeks prior to registration
* Immunocompromised patients and patients with known immunodeficiency; or receiving systemic steroid therapy or any other immunosuppressive therapy =< 7 days prior to registration; NOTE: inhaled steroids and low-dose corticosteroids are allowed
* History of active tuberculosis (TB), human immunodeficiency virus (HIV), active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) and/or active hepatitis C infection (e.g. hepatitis C virus [HCV] ribonucleic acid [RNA] qualitative is detected)
* Received a live vaccine =< 30 days prior to registration; NOTE: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines, and are not allowed
* Hypersensitivity to pembrolizumab, binimetinib, or any excipients of either drug
* Prior anti-cancer therapy with a monoclonal antibody (mAb) =< 4 weeks prior to registration OR failure to recover (to =< grade 1) from adverse events (AE) attributable to agents received > 4 weeks prior to registration
* Prior therapy including chemotherapy, targeted small molecule therapy or radiation therapy =< 2 weeks prior to registration OR failure to recover (to =< grade 1 or to baseline) from adverse events (AE) attributable to agents received > 4 weeks prior to registration; NOTE: exception for neuropathy =< grade 2, which is allowed
* Any active central nervous system (CNS) lesion (i.e., those with radiographically unstable, symptomatic lesions) and/or leptomeningeal metastases; NOTE: patients treated with stereotactic radiotherapy or surgery are eligible if no evidence of CNS disease progression >= 4 weeks and patients must be off corticosteroid therapy for >= 3 weeks; NOTE: carcinomatous meningitis is excluded regardless of clinical stability
* Active autoimmune disease requiring systemic treatment in the past 2 years (i.e. use of disease modifying agents, corticosteroids or immunosuppressive drugs); NOTE: replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Known history of, or any evidence of active, non-infectious pneumonitis
* Active infection requiring systemic therapy
* Known history of acute or chronic pancreatitis
* History of or current evidence of retinal vein occlusion (RVO) or predisposing factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
* History of retinal degenerative disease
* History of Gilbert's syndrome
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: adequately treated non-melanotic skin cancer (adequate wound healing is required prior to study entry) or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior solid tumor malignancy, it must have been treated curatively with no evidence of recurrence =< 3 years prior to registration
* Impaired cardiovascular function or clinically specific cardiovascular disease including any of the following:

  * History of acute coronary syndromes (including myocardial infarction unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) =< 6 months; OR
  * Symptomatic chronic heart failure history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality < 6 months prior to screening; except atrial fibrillation and paroxysmal supraventricular tachycardia
* Uncontrolled arterial hypertension defined as persistent elevation of systolic blood pressure >= 150 mmHg or diastolic blood pressure >= 100 mmHg despite medical treatment
* History of neuromuscular disorders that are associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Planning to embark on a new strenuous exercise regimen after first dose of study treatment; NOTE: muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on binimetinib treatment
* Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection); NOTE: gastric bypass is allowed
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/psychological issues, etc.
* Major surgery =< 3 weeks prior to registration or failure to adequately recover from surgery
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study
* RETREATMENT REGISTRATION: Received any type anti-cancer treatment since the last dose of pembrolizumab
* RETREATMENT REGISTRATION: History or current evidence of any condition, therapy, or laboratory abnormality that might interfere with subject's participation for the full duration of the trial or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 0: Patients receive 45mg binimetinib PO BID on days 1-14 of cycle 1 and on days 1-21 of cycle 2 and subsequent cycles. Beginning cycle 2, patients also receive 200mg pembrolizumab IV over 30 minutes on day 1. Cycle 1 equals 14 days. Cycles 2 and beyond repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level -1; Phase 2: Patients receive 30mg binimetinib PO BID on days 1-14 of cycle 1 and on days 1-21 of cycle 2 and subsequent cycles. Beginning cycle 2, patients also receive 200mg pembrolizumab IV over 30 minutes on day 1. Cycle 1 equals 14 days. Cycles 2 and beyond repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Phase 1
Arm/Group | Phase 1 Dose Level 0 | Phase 1 Dose Level -1 | Phase 2
Started | 5 | 8 | 0
Completed | 3 | 6 | 0
Not Completed | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Period: Phase 2
Arm/Group | Phase 1 Dose Level 0 | Phase 1 Dose Level -1 | Phase 2
Started | 0 | 8 | 10
Completed | 0 | 8 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 0 | Phase 1 Dose Level -1 | Phase 2 | Total
Number analyzed (Participants) | 5 | 8 | 10 | 23
Age, Continuous [Median (Full Range); unit: years] | 63 [57 to 69] | 62 [37 to 77] | 54.5 [40 to 65] | 58 [37 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 10 | 23
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 10 | 21
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 1 | 8
  White | 1 | 4 | 7 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Pembrolizumab in Combination With Binimetinib Using the Standard 3+3 Design (Phase I)
Description: Will be assessed by Common Terminology Criteria for Adverse Events version 4.0. Safety/adverse events data will be tabulated, including adverse events of all grades.
Time Frame: 35 days
Population: All patients treated per protocol and evaluated for dose limiting toxicities.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 0 | Phase 1 Dose Level -1
Number analyzed (Participants) | 3 | 6
Participants
  Experienced Dose Limiting Toxicity | 2 | 0
  No Dose Limiting toxicity | 1 | 6

2. Primary Outcome: Objective Response Rate (ORR) as (Phase II)
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST). Will utilize Simon's Two-Stage Optimal Design to test the null hypothesis. Will be estimated using the approach of Jung and Kim. The 90% lower confidence bound will be calculated using the approach of Koyama and Chen. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 3 years
Population: Phase 1 dose level -1 patients are included with phase 2 patients in order to increase the strength of analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Phase 2
Number analyzed (Participants) | 18
Proportion of participants | .304 [.122 to .473]

3. Secondary Outcome: ORR by Immune-related RECIST Criteria (irRECIST)
Description: The Overall Response Rate, ORR, is defined as the proportion of patients with a response per irRECIST. It will be estimated as a binomial proportion with a 2-sided 95% confidence intervals. Baseline tumor infiltrating lymphocyte (TILs) and percent change in TILs from baseline will be summarized. Logistic regression models will be used to assess the correlation between these biomarkers and ORR in order to assess their prognostic significance.
Time Frame: Up to 3 years
Population: Only patients treated at the maximum tolerated dose level 0f -1 are evaluable for this phase 2 response analysis. Phase 1 dose level -1 patients and Phase 2 dose level -1 patients were combined for this analysis. Patients treated on other dose levels explored during the phase 1 portion, such as dose level 0, are excluded.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- All Dose Level -1: Patients receive 30mg binimetinib PO BID on days 1-14 of cycle 1 and on days 1-21 of cycle 2 and subsequent cycles. Beginning cycle 2, patients also receive 200mg pembrolizumab IV over 30 minutes on day 1. Cycle 1 equals 14 days. Cycles 2 and beyond repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Dose Level -1
Number analyzed (Participants) | 18
proportion of participants | 0.278 [0.097 to 0.535]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Patients who are alive (including those lost to follow-up) at the time of data analysis will be censored at the last known alive date. A Kaplan-Meier curve will be used to summarize the PFS experience of this patient cohort. Cox Proportional Hazard models will be used to assess baseline TILs and percent change in TILs from baseline and their correlation with PFS. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: The time from study enrollment to date of progression, assessed up to 3 years
Population: All treated and evaluable patients were analyzed by dose level.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Dose Level 0: Patients receive 45mg binimetinib PO BID on days 1-14 of cycle 1 and on days 1-21 of cycle 2 and subsequent cycles. Beginning cycle 2, patients also receive 200mg pembrolizumab IV over 30 minutes on day 1. Cycle 1 equals 14 days. Cycles 2 and beyond repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Dose Level 0 | All Dose Level -1
Number analyzed (Participants) | 4 | 18
Months | 2.43 [0.49 to NA] — Due to lack of events the upper limit was not reached | 7.92 [3.88 to NA] — Due to lack of events the upper limit was not reached

5. Secondary Outcome: Overall Survival (OS)
Description: Patients who are alive (including those lost to follow-up) at the time of data analysis will be censored at the last known alive date. A Kaplan-Meier curve will be used to summarize the OS experience of this patient cohort. Cox Proportional Hazard models will be used to assess baseline TILs and percent change in TILs from baseline and their correlation with OS.
Time Frame: The time from study enrollment to death attributable to any cause, assessed up to 3 years
Population: All treated and evaluable patients were analyzed by dose level.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Dose Level 0 | All Dose Level -1
Number analyzed (Participants) | 4 | 18
Months | 7.03 [0.49 to NA] — Due to lack of events the upper limit was not reached | 33.18 [11.24 to NA] — Due to lack of events the upper limit was not reached

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 3 years and mortality was followed for 4.5 years
Description: One Phase 1 Dose Level 0 patient was never treated or assessed for adverse events
Arm/Group | Phase 1 Dose Level 0 | Phase 1 Dose Level -1 | Phase 2
All-Cause Mortality (participants affected / at risk) | 5/5 | 4/8 | 7/10
Serious Adverse Events (participants affected / at risk) | 1/4 | 3/8 | 5/10
Other Adverse Events (participants affected / at risk) | 3/4 | 8/8 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 0 (N=4) | Phase 1 Dose Level -1 (N=8) | Phase 2 (N=10)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 0 (N=4) | Phase 1 Dose Level -1 (N=8) | Phase 2 (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 5 (34) | 8 (27)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (5) | 6 (20) | 9 (48)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 2 (11) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (4)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (4) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (3) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (3)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (5) | 6 (13)
Blurred vision (Eye disorders) | 0 (0) | 2 (31) | 2 (3)
Cataract (Eye disorders) | 0 (0) | 1 (33) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 3 (26) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (3) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital edema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (7) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (3) | 4 (54) | 6 (20)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 4 (15) | 7 (20)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (15) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (33) | 2 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 4 (43) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (4) | 7 (15) | 7 (29)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 4 (12)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 5 (40) | 4 (17)
Fatigue (General disorders) | 2 (5) | 7 (86) | 9 (42)
Fever (General disorders) | 0 (0) | 1 (1) | 2 (2)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (31) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (1) | 1 (5)
Bladder infection (Infections and infestations) | 0 (0) | 1 (6) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Corneal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 3 (6) | 3 (10)
Sinusitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (11) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (19) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 0 (0)
Activated partial throm time prolonged (Investigations) | 0 (0) | 3 (15) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 6 (12)
Alkaline phosphatase increased (Investigations) | 1 (2) | 2 (13) | 6 (23)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 3 (7) | 9 (31)
CPK increased (Investigations) | 2 (6) | 4 (36) | 6 (28)
Cardiac troponin T increased (Investigations) | 0 (0) | 6 (87) | 7 (22)
Creatinine increased (Investigations) | 0 (0) | 2 (5) | 2 (13)
ECG QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (18) | 2 (10)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 5 (7)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (16) | 2 (4)
Platelet count decreased (Investigations) | 0 (0) | 2 (30) | 2 (4)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (5)
White blood cell decreased (Investigations) | 0 (0) | 1 (9) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (23) | 3 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (10) | 5 (11)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (8) | 3 (6)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (13) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (40) | 1 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (8)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (14) | 3 (17)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (32) | 2 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (31) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (7)
Ataxia (Nervous system disorders) | 0 (0) | 1 (30) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (5) | 3 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (37) | 3 (14)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 1 (6) | 1 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (4) | 7 (96) | 4 (13)
Presyncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (22) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (4) | 1 (2)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 2 (16) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 2 (8) | 1 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (17) | 3 (7)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 2 (8) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (8) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (5) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (3)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (4)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 1 (4)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (14) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (21) | 1 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (19) | 5 (6)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (14) | 1 (6)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (20) | 4 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (22) | 3 (6)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (12) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (27) | 4 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (6) | 3 (5) | 4 (22)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 7 (21)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (16) | 5 (9)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Hot flashes (Vascular disorders) | 0 (0) | 2 (10) | 1 (8)
Hypertension (Vascular disorders) | 0 (0) | 5 (31) | 3 (15)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 2 (44) | 3 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT03106415/Prot_SAP_000.pdf